CLINICAL TRIAL: NCT04739501
Title: Trans-arterial Chemoembolization in Patients With Hepatocellular Carcinoma
Brief Title: Trans-arterial Chemoembolization in Patients With Hepatocellular Carcinoma: A Study of Different Outcomes and Their Predictive Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Mahran Mohammed Ahmed, resident of tropical medicine, Assiut University
Other Study IDs: 0987654321
Record Dates: First submitted 2020-03-25; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 35 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TACE in HCC group 1: the patient did undergo tace
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — Trans-arterial chemoembolization in patients with hepatocellular carcinoma

SUMMARY:
Radiological response after trans arterial chemoembolization (TACE) is classified according to Modified Response Evaluation Criteria in Solid Tumors (mRECIST) to: complete response (CR) (disappearance of arterial enhancement), partial response (PR) ( at least a 30% decrease in the sum of diameters of viable enhancement), progressive disease (PD) (an increase of at least 20% in the sum of the diameters of viable enhancement, or appearance of new lesions), and stable disease (any cases that do not qualify for either partial response or progressive disease

DETAILED DESCRIPTION:
POST-TACE response of treatment for cases of hepatocellular cancer

ELIGIBILITY:
Inclusion Criteria:

Clinical history and examination with special stress on symptoms and signs of chronic liver disease with or without evidence of hepatic decompensation e.g. the presence of ascites and with or without evidence of complications e.g. jaundice spider naevi, bleeding varices, ascites, and lower limb edema.

Laboratory findings in the form of raised bilirubin and liver enzymes, impaired coagulation profile, and/or low serum albumin.

Abdominal ultrasonography revealing liver cirrhosis (coarse echopattern, attenuated hepatic veins, irregular outlines, hypertrophy of caudate lobe and/or shrunken liver, presence of focal hepatic) and presence of splenomegaly, ascites, or portal vein thrombosis (PVT).

Exclusion Criteria:

A patient who had surgical resection or liver transplantation Patients refuse to participate Hepatic focal lesion other than HCC

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HCC with TACE
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Post_TACE hepatic cell failure | 1 year
  Frequency of liver cell failure in form of jaundice , coagulopathy and encephalopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No